CLINICAL TRIAL: NCT04517851
Title: A Pilot Study of the Anti-SLAMF7 Monoclonal Antibody, Elotuzumab, in Patients With Myelofibrosis
Brief Title: Elotuzumab for the Treatment of JAK2-Mutated Myelofibrosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0522; NCI-2020-05712 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0522 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis Transformation in Essential Thrombocythemia; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Primary Myelofibrosis
MeSH Terms: conditions — Polycythemia Vera; Primary Myelofibrosis | interventions — elotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (elotuzumab) (Experimental): Patients receive elotuzumab IV over 1-4 hours on days 1, 8, 15, and 22 of cycles 1-2. Beginning in cycle 3, patients receive elotuzumab IV over 1-4 hours on day 1. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Elotuzumab; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Elotuzumab — Given IV
  Other Names: BMS-901608; Empliciti; HuLuc-63; HuLuc63; PDL-063; PDL063
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial investigates how well elotuzumab works in treating patients with JAK2-mutated myelofibrosis. Elotuzumab may help to control myelofibrosis and/or help to improve blood cell count and bone marrow function.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To obtain preliminary evidence of the efficacy of elotuzumab in patients with myelofibrosis (MF) by estimating the rate of overall response by International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) 2013 criteria.

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of elotuzumab in patients with MF.

II. To assess for improvements in cytopenias and bone marrow fibrosis grade, splenomegaly and disease-related symptoms.

III. To determine the duration of objective responses, if any, to elotuzumab. IV. To determine the time to next treatment.

EXPLORATORY OBJECTIVES:

I. To assess the proportion of circulating monocytes expressing the target of elotuzumab, SLAMF7, and any correlation of the same to the mutant JAK2 allele burden.

II. To assess baseline levels of IL-1Ralpha and other cytokines and the effects of elotuzumab, if any, on these over time.

III. To examine the effects of elotuzumab on fibrocyte count and differentiation, both in vitro and in vivo.

IV. To assess clonal evolution, if any, in MF patients on elotuzumab treatment.

OUTLINE:

Patients receive elotuzumab intravenously (IV) over 1-4 hours on days 1, 8, 15, and 22 of cycles 1-2. Beginning in cycle 3, patients receive elotuzumab IV over 1-4 hours on day 1. Treatment repeats every 28 days for up to 36 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Adults with JAK2 V617F+ primary myelofibrosis (PMF) or post-polycythemia vera (PV)/essential thrombocythemia myelofibrosis (ET-MF) who require treatment and have intermediate or higher risk disease (as assessed by the International Prognostic Scoring System for Myelodysplastic Syndrome [IPSS], Dynamic International Prognostic Scoring System [DIPSS], DIPSS-plus, Mutation-Enhanced Prognostic System for Transplant Age Patients with Primary Myelofibrosis [MIPSS70], MIPSS70-plus version [v] 2.0, or MYelofibrosis SECondary to PV and ET-Prognostic Model [MYSEC-PM]). The MYSEC-PM is to only be used for patients with post-PV/ET MF
* Patients must not be candidates for JAK inhibitor therapy in the opinion of the treating physician
* Bone marrow (BM) fibrosis grade 2 or 3 according to the European classification
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 (Karnofsky performance status >= 60%)
* Absolute neutrophil count >= 0.5 x 10^9/L
* Direct bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless felt to be due to liver involvement by MF/extramedullary hematopoiesis, in which case =< 5 x institutional upper limit of normal is permissible
* Creatinine =< 2 x institutional upper limit of normal OR creatinine clearance >= 30 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation until 6 months after the last administration of elotuzumab. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Women of child-bearing potential must have a negative pregnancy test. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after the last administration of elotuzumab

Exclusion Criteria:

* Splenic irradiation within the preceding 4 months
* Chemotherapy (other than hydroxyurea), interferons, IMiDs, danazol or other androgens, erythroid stimulating agents, or other MF-directed commercially available agents within 4 weeks prior to entering the study or those who have not recovered to baseline from adverse events due to agents administered more than 4 weeks earlier
* Other investigational agents within 4 half-lives prior to study entry
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to elotuzumab
* Patients with known central nervous system (CNS) involvement
* Prior allogeneic hematopoietic cell transplantation (allo-HCT) for MF
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known pregnancy or lactation
* Known human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response (OR) | Up to completion of cycle 36 (1 cycle is 28 days)
  OR is defined as CR (complete response) +PR (partial response) + CI (clinical improvement), where CI includes clinical improvements in anemia, splenomegaly and/or symptoms. Will estimate the OR rate, along with the exact 95% confidence interval.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post-treatment
  The method of Thall, Simon and Estey will be used to monitor for safety. The severity of the toxicities will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 whenever possible. Will follow standard reporting guidelines for adverse events. Safety data will be summarized by category, severity and frequency.
Duration of response | Up to 5 years
  The Kaplan-Meier method will be used to estimate the duration of response where median and 95% confidence interval will be reported.
Time to next treatment | Up to 5 years
  The Kaplan-Meier method will be used to estimate the time to next treatment where median and 95% confidence interval will be reported.
Rates of complete response | Up to 5 years
Rates of partial response | Up to 5 years
Rates of clinical improvement | Up to 5 years
Platelet response rate | Up to 5 years
Changes in bone marrow fibrosis grade | Baseline up to 5 years
  Will be assessed according to European classification.

OTHER OUTCOMES:
Biomarker analysis | Up to 5 years
  Fisher's exact test will be used to assess the associations between biomarker expression (high versus low) and outcomes. Wilcoxon singed rank test will be applied to assess the change of biomarkers from baseline.
Percentage of circulating SLAMF7high/CD16neg monocytes | Baseline and over time up to 5 years
Serum IL-1Ralpha levels | Baseline and over time up to 5 years
JAK2V617F allele burden in the bone marrow or blood | Baseline and over time up to 5 years
Myeloid mutation panel (81-gene next generation sequencing panel) on serial bone marrow aspirates | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prithviraj Bose, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org